CLINICAL TRIAL: NCT05626608
Title: Neuromodulation électrique Continue du Globus Pallidus Dans la Maladie de Parkinson Par l'électrode Directionnelle CARTESIA™
Brief Title: Continuous Electrical Neuromodulation of the Globus Pallidus Intern in Parkinson's Disease by the Directional Electrode CARTESIA™
Acronym: NEC-Parkinson
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: RECHMPL20_0466
Record Dates: First submitted 2022-11-07; First posted 2022-11-25 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Parkinson Disease
Keywords: Deep Brain Stimulation (DBS); Directional Stimulation; Subthalamic Nucleus (STN); Imaging Based Targeting; Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Two of the 4 investigators will not be aware of the stimulation modality programmed in the patient.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Directional (Experimental): Directional stimulation of the subthalamic nucleus in the treatment of Parkinson's disease using Boston Cartesia(TM) electrodes
  Interventions: Device: Stimulation in directional mode
- Conventional ring (Monopolar and Bipolar) (Active Comparator): Unilateral or bilateral subthalamic nucleus stimulation in the treatment of Parkinson's disease using Boston Cartesia(TM) electrodes
  Interventions: Device: Classical ring stimulation

INTERVENTIONS:
Device: Classical ring stimulation — Unilateral or bilateral subthalamic nucleus stimulation in the treatment of Parkinson's disease using Boston Cartesia(TM) electrodes
  Arms: Conventional ring (Monopolar and Bipolar)
Device: Stimulation in directional mode — Directional stimulation of the subthalamic nucleus in the treatment of Parkinson's disease using Boston Cartesia(TM) electrodes
  Arms: Directional

SUMMARY:
Many patients have benefited from the implantation of brain stimulation electrodes for the treatment of various motor signs of Parkinson's disease in the phase of motor fluctuations. This technique has significantly improved the motor symptomatology of Parkinson's disease and the dyskinesias induced by pharmacological treatment. Technological advances in the field of deep brain stimulation (DBS) could improve the benefit of this therapeutic tool. therapeutic tool. While using directional electrodes, it remains possible to program the stimulation in conventional ring mode.

DETAILED DESCRIPTION:
Idiopathic Parkinson's disease represents the second degenerative disease after Alzheimer's disease, with progressive motor and non-motor symptoms, affecting the dopaminergic system (at the origin of the cardinal symptoms) and the other systems, cholinergic, noradrenergic and serotonergic (responsible for the dopa-resistant symptoms). The functional repercussions are important and a source of handicap in the more advanced phases of the disease. Many patients have benefited from the implantation of deep brain stimulation (DBS) electrodes, associated with dopaminergic replacement therapy, for the treatment of various motor signs of Parkinson's disease in the phase of motor fluctuations.

It is an advanced symptomatic therapy that does not prevent the progression of the disease. DBS is intended for Parkinson's patients in the phase of motor fluctuations. The aim of this treatment is to complement the therapeutic effect of pharmacological treatments that patients will have to continue as well as to compensate for certain effects induced by the drugs. The effectiveness of DBS therapy may decrease over time, especially in the context of a progressive pathology, and requires a change of batteries after several years (4 to 15 years, depending on the type of neurostimulator, non-rechargeable or rechargeable).

Beyond these constraints, this adaptable therapy has significantly improved the motor symptomatology of Parkinson's disease and the dyskinesias induced by pharmacological treatment. Technological advances in DBS could improve the therapeutic benefit of this technique and limit its side effects (dysarthria, hypophonia, oculomotor disorders, muscular contractions induced by the diffusion of the current), by using different modalities of brain stimulation. Implantation of Boston Scientific Cartesia™ directional electrodes for Parkinson's patients who are candidates for deep brain stimulation of the subthalamic nucleus (STN) would allow reorientation and variation of the volume of the stimulated structure, which could improve therapeutic performance, by stimulating key target volumes for obtaining the clinical effect, limiting side effects by diffusion of the current on neighboring structures. While using directional electrodes, it remains possible to program the stimulation in ring mode, conventional stimulation modality, in monopolar or bipolar.

The hypothesis is that the efficacy of DBS in directional mode will be more effective on the motor signs of Parkinson's disease compared to omnidirectional stimulation and bipolar mode, with a better tolerance profile (fewer side effects).

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of bilateral idiopathic Parkinson's disease according to the British Brain Bank criteria (bradykinesia and rigidity or resting tremor)
* Parkinson's disease that has been evolving for several years (>4 years)
* Persistence of a good sensitivity to L-Dopa, essential criterion in the selection, except for tremor (Improvement in Parkinson's disease symptoms of at least 30% measured on the UPDRS, section III)
* A UPDRS (Unified Parkinson Disease Rating Scale) part III motor score >25 under MEDOFF conditions
* Patient with tremor not controlled́ by treatment and which represents the bulk of the symptomatology. Patient will require stable treatment throughout the study.
* Patient with major motor fluctuations with prolonged blocking and/or dyskinesias
* Be a candidate for PCS and bilateral electrode implantation in the STN.
* A Hoehn and Yahr scale score ≤ 2.5 under best MED-ON conditions
* A UPDRS section II activities of daily living score > 6
* Patient without comorbidities that do not allow the patient to undergo general anesthesia general anesthesia or a neurosurgical procedure or interfering with the follow-up required by the protocol

Exclusion Criteria:

* Characterized depressive episode (BDI>25) (depressive episodes prior to inclusion and completed at the time of inclusion will not be considered as a non-inclusion criterion)
* Psychotic episodes (Brief Psychiatric Rating Scale, BPRS) (mild hallucinations or acute psychotic episodes preceding the screening and inclusion period and completed at the time of inclusion will not be considered as non-inclusion criteria)
* Dementia (Mattis DRS score <125)
* Contraindication to general anesthesia
* Absolute MRI contraindications: Pacemaker or neurosensory stimulator or implantable defibrillator; Cochlear implants; Ocular or cerebral ferromagnetic foreign bodies close to nerve structures
* Relative MRI contraindications: Metallic prostheses, especially orthodontic braces; Patient agitation; Pregnant women; Ventriculoperitoneal neurosurgical shunt valves; Tattoos containing iron particles
* Contraindication revealed by abnormal cerebral MRI (after-effects of stroke, vascular malformations, major cerebral atrophy)
* Serious intercurrent pathology
* Surgical contraindication
* Pregnancy in progress or planned during the study period, Pregnant or breastfeeding women or women in a state of procreation without contraception Women who are pregnant or breastfeeding or in a state of procreation without effective contraception
* Impossibility or refusal of regular follow-up of at least 30 months
* Participation in other interventional research
* Adult protected by law or patient under guardianship or curatorship
* Patient unable to use the remote control and charging system properly or who does not have a person who can assist them in this process
* Failure to obtain written informed consent after a period of reflection
* Not being affiliated to a French social security system or being a beneficiary of such a system

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2023-04-28 (Actual); Primary Completion 2026-10-28 (Estimated); Study Completion 2026-10-28 (Estimated)

PRIMARY OUTCOMES:
Comparison of motor scores | 12 months
  Comparison of motor scores between classical ring, monopolar or bipolar stimulation and stimulation in directional mode thanks to the part III of the UPDRS (Unified Parkinson Disease Rating Scale). The total score ranges from 0 (no disability) to 60 (total disability).

SECONDARY OUTCOMES:
Evaluation of patient acceptability for a stimulation modality | 12 months
  Evaluate for which programming modality(ies) the percentage of patients is most important
Evaluation of the tolerance of different types of stimulation | 12 months
  Collection of induced side effects (dysarthria, hypertonia, oculomotor disorders)
Evaluation of the clinical effects of programming functions | 12 months
  The additional percentage improvement in clinical scores versus directional stimulation without the use of the focus function at each visit.
Evaluation of clinical effects of Directional programming mode | 12 months
  the clinical effects of different directions on motor symptoms will be evaluated and compared to the ring, monopolar and bipolar stimulation modalities, for the two plots evaluated as being the most effective in controlling motor signs and with the widest therapeutic window. The evaluation will be made thanks to the part III of the UPDRS (Unified Parkinson Disease Rating Scale). The total score ranges from 0 (no disability) to 60 (total disability).

CONTACTS AND LOCATIONS:
Overall Officials: Gaëtan POULEN, PD, Study Director — CHU de Montpellier
Locations (1):
- Centre Hospitalier Uniersitaire de Montpellier, Montpellier, France, France